CLINICAL TRIAL: NCT05799950
Title: A Real-World Evidence (RWE) Long-Term Follow-Up Study to Assess Outcomes of Alcon Monofocal Intraocular Lenses
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: ILB609-N001
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Aphakia
Keywords: Intraocular lens; Cataract
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- AcrySof single-piece IOL: Pseudophakic subjects previously implanted with an AcrySof single-piece IOL
  Interventions: Device: AcrySof single-piece IOL
- AcrySof multi-piece IOL: Pseudophakic subjects previously implanted with an AcrySof multi-piece IOL
  Interventions: Device: AcrySof multi-piece IOL

INTERVENTIONS:
Device: AcrySof single-piece IOL — Acrylic single-piece intraocular lens placed in the capsular bag in the posterior chamber of the eye during cataract surgery as a replacement for the natural crystalline lens.
  Other Names: Models SN60WF, ACU0T0, SN6AT2, SN6AT3, SN6AT4, SN6AT5, SN6AT6, SN6AT7, SN6AT8, SN6AT9, SA6AT2, SA6AT3, SA6AT4, SA6AT5, SA6AT6, SA6AT7, SA6AT8, SA6AT9
  Groups: AcrySof single-piece IOL
Device: AcrySof multi-piece IOL — Acrylic multi-piece intraocular lens placed in the capsular bag in the posterior chamber of the eye during cataract surgery as a replacement for the natural crystalline lens.
  Other Names: Models MN50BM, MA60AC, MA60MA
  Groups: AcrySof multi-piece IOL

SUMMARY:
The purpose of this post-market clinical follow-up (PMCF) study is to describe the long-term safety and performance of AcrySof Single-Piece and AcrySof Multi-Piece monofocal intraocular lenses (IOLs).

DETAILED DESCRIPTION:
The study includes a retrospective chart review for pre-operative, operative, and post-operative data collection, and a prospective, standard-of-care visit to collect study endpoints.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject is implanted with one of the study IOL models between 3 and 5 years previously.
* Subject follow-up is expected to be possible during the duration of the study.
* Subject or legally authorized representative must be able to understand and sign the IRB/EC approved Informed Consent form. Minor subjects will complete an Assent Form.
* Documented medical history and required pre-operative baseline information is available for retrospective data collection.

Key Exclusion Criteria:

* Subject is participating in a separate investigational drug or device study.
* Pregnancy at the time of enrollment.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from clinical sites in the United States and Canada.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Mean monocular best corrected distance visual acuity (BCDVA) | Up to 3 to 5 years post operative
  Retrospectively, the subject's medical records will be reviewed for assessments of BCDVA. Prospectively, visual acuity will be assessed for each eye individually with correction in place using letter charts placed at a distance of 6 meters (or 4 meters adjusted for infinity) from the subject. BCDVA will be reported in logarithm minimum angle of resolution (logMAR), where a logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight) and lower logMAR values indicate better visual acuity.
Rate of protocol-specified ocular adverse events | Up to 3 to 5 years post operative
  The subject's medical records will be reviewed for medical conditions. Medical conditions that started after initial exposure to the study model IOLs will be captured as adverse events. The following adverse events are pre-specified for this outcome measure:
  * Cystoid macular edema (CME)
  * Hypopyon
  * Endophthalmitis
  * Lens dislocation
  * Pupillary block
  * Retinal detachment
  * Secondary surgical interventions

SECONDARY OUTCOMES:
Mean manifest refraction - Sphere | Up to 3-5 years postoperative
  Retrospectively, the subject's medical records will be reviewed for manifest refraction assessments. Prospectively, the subject will be manually refracted to his/her best correction using a phoropter. The spherical component will be measured in diopters.
Mean manifest refraction - Cylinder | Up to 3-5 years postoperative
  Retrospectively, the subject's medical records will be reviewed for manifest refraction assessments. Prospectively, the subject will be manually refracted to his/her best correction using a phoropter. The cylindrical component will be measured in diopters.
Mean manifest refraction - Axis | Up to 3-5 years postoperative
  Retrospectively, the subject's medical records will be reviewed for manifest refraction assessments. Prospectively, the subject will be manually refracted to his/her best correction using a phoropter. The axial component will be measured in degrees.
Manifest refraction spherical equivalent (MRSE) | Up to 3-5 years postoperative
  Retrospectively, the subject's medical records will be reviewed for manifest refraction assessments. Prospectively, the subject will be manually refracted to his/her best correction using a phoropter. MRSE will be calculated as [Sphere minus (cylinder divided by 2)] and reported in diopters.
Mean monocular uncorrected distance visual acuity (UCDVA) | Up to 3-5 years postoperative
  Visual acuity will be assessed for each eye individually with no correction in place using letter charts placed at a distance of 6 meters (or 4 meters adjusted for infinity) from the subject. UCDVA will be measured in logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with lower logMAR values indicating better visual acuity.
Rate of additional adverse events - Ocular | Up to 3-5 years postoperative
  The subject's medical records will be reviewed for medical conditions. Medical conditions that started after initial exposure to the study model IOLs will be captured as adverse events. This outcome measure will include all ocular adverse events other than the protocol-specified adverse events.
Rate of device deficiencies | Up to 3-5 years postoperative
  The subject's medical records will be reviewed for device deficiencies. Examples of device deficiencies include the following:
  * Failure to meet product specifications (e.g., incorrect IOL power);
  * IOL defect;
  * Broken IOL optic;
  * Broken IOL haptic; Scratched IOL optic;
  * Unsealed device packaging;
  * Suspected product contamination;
  * Lack of performance. A device deficiency may or may not be associated with subject harm.
Rate of posterior capsulotomies | Up to 3-5 years postoperative
  Posterior capsulotomy is surgery performed on the back side of the capsular bag in the eye. A laser is used to make an opening in the cloudy capsule to allow light to pass through again for clear vision. The subject's medical records will be reviewed for the occurrence of posterior capsulotomy.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Lead, Surgical, Study Director — Alcon Research, LLC
Locations (7):
- United States (6):
  - Velvet Clinical Research, Burbank, California
  - Levenson Eye Associates, Jacksonville, Florida
  - Virdi Eye Clinic, Rock Island, Illinois
  - SightMD, Babylon, New York
  - Texan Eye, Austin, Texas
  - Chu Eye Institute, Fort Worth, Texas
- Centro Oftalmologico Metropolitano, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No